CLINICAL TRIAL: NCT06414811
Title: Prediction of TAPSE/PASP Ratio for Hypotension Due to General Anesthesia Induction
Brief Title: Tapse/Pasp General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, ASS. PROF. DR, Aydin Adnan Menderes University
Other Study IDs: 2024-44
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-05

CONDITIONS: Hypotension
Keywords: TAPSE; PASP; GENERAL ANESTHESİA
MeSH Terms: conditions — Hypotension | interventions — Hypotension, Controlled; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypotension: Patients with a 30% decrease in SBP from baseline and a decrease in MAP below 65 mmHg in the first 10 minutes after anesthesia induction will be considered to have hypotension.
  Interventions: Other: HYPOTENSİON
- none hypotension: Patients who do not have a 30% decrease from the baseline in SBP and a decrease in MAP below 65 mmHg in the first 10 minutes after anesthesia induction will be considered as not having hypotension.

INTERVENTIONS:
Other: HYPOTENSİON — MAP below 55 mmHg or long-term (2 minutes or more) hypotensive attacks will be treated with ephedrine 0.1mg/kg.
  Other Names: TREATMENT
  Groups: Hypotension

SUMMARY:
TAPSE, one of the methods for evaluating right ventricular systolic function; It is a bar parameter that can easily measure apex-basal shortening and provides specific information about global RV function. TAPSE/PASP can be calculated as load-independent parameters to evaluate RV function. Because RV function is sensitive to change in afterload, known as the RV-pulmonary circulation (PC) connection.

This study aims to identify patients who are candidates for hypotensive events due to general anesthesia in a hemodynamically stable population.

DETAILED DESCRIPTION:
TAPSE, one of the methods for evaluating right ventricular systolic function; It is a bar parameter that can easily measure apex-basal shortening and provides specific information about global RV function. TAPSE/PASP can be calculated as load-independent parameters to evaluate RV function. Because RV function is sensitive to change in afterload, known as the RV-pulmonary circulation (PC) connection.

This study aims to identify patients who are candidates for hypotensive events due to general anesthesia in a hemodynamically stable population.

Patients will be measured by transthoracic echocardiography in the preoperative period, 15-30 minutes before induction.

Basal hemodynamic parameters and non-invasive and/or hemodynamic values will be recorded every two minutes after induction until surgical incision.Patients with a 30% decrease in SBP from the baseline and a decrease in MAP below 65 mmHg in the first 10 minutes after anesthesia induction will be considered to have hypotension. Patients will be divided into 2 groups: 'with' and 'without' hypotension.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. 18-75 years old
3. ASA Physical Status 1-3;
4. Patients planned for surgery

Exclusion Criteria:

1. The patient is pregnant
2. After cardiac surgery
3. Severe pulmonary hypertension
4. Severe valve disease
5. Hypertrophic or dilated cardiomyopathy
6. Presence of acute myocardial infarction
7. Patients with severe visual or hearing impairment/disability
8. ASA physical status IV or V
9. Ischemic heart disease, conduction disorder.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ASA1-3 patients aged 18-75 who will undergo elective surgery
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
1. tension | 4-5 hours]
  Intraoperative systolic arterial tension, diastolic arterial tension and mean arterial tension will be taken and recorded for the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Ferdi Gülaştı, Aydin, Turkey (Türkiye)